CLINICAL TRIAL: NCT07304830
Title: The Effects of the PsyPills App on Emotion Regulation and Risk Behaviors in Emerging Adults: A Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Oana David, Professor PhD, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PsyPills-Risk-Behaviors
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Emotion Regulation Difficulties; Risky Behaviors (Substance Use, Risky Sexual Behavior, Self-harm, Aggression, Disordered Eating)
MeSH Terms: conditions — Substance-Related Disorders; Self-Injurious Behavior; Aggression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PsyPills (Experimental): A self-guided mobile intervention based on Rational-Emotive and Behavioral Therapy (REBT) principles and the Just-in-Time Adaptive Intervention (JITAI) framework. Provides short, adaptive "psychological pills" - personalized cognitive restructuring exercises aimed at identifying and replacing irrational beliefs, reducing dysfunctional emotionality, and improving emotion regulation.
  Interventions: Behavioral: PsyPills
- MoodWheel (Active Comparator): The active control condition involves using the MoodWheel app, designed for emotional self-monitoring without therapeutic content. Participants label and track their emotional states, but the app does not provide cognitive restructuring, feedback, or intervention elements.
  Interventions: Behavioral: MoodWheel

INTERVENTIONS:
Behavioral: PsyPills — A self-guided mobile intervention based on Rational-Emotive and Behavioral Therapy (REBT) principles and the Just-in-Time Adaptive Intervention (JITAI) framework. Provides short, adaptive "psychological pills" - personalized cognitive restructuring exercises aimed at identifying and replacing irrational beliefs, reducing dysfunctional emotionality, and improving emotion regulation.
  Arms: PsyPills
Behavioral: MoodWheel — The active control condition involves using the MoodWheel app, designed for emotional self-monitoring without therapeutic content. Participants label and track their emotional states, but the app does not provide cognitive restructuring, feedback, or intervention elements.
  Arms: MoodWheel

SUMMARY:
This study aims to investigate the effects of the PsyPills mobile application on improving emotion regulation and reducing risk behaviors among emerging adults. PsyPills is a self-guided psychological intervention based on Rational-Emotive and Behavioral Therapy (REBT) principles and the Just-in-Time Adaptive Intervention (JITAI) framework. The app provides short, contextually adaptive "psychological pills," or cognitive restructuring exercises, designed to help users replace irrational beliefs with rational alternatives in moments of emotional distress. The study will compare PsyPills app with an active control condition using the MoodWheel app, which supports emotional monitoring without therapeutic content.

DETAILED DESCRIPTION:
The research design will be a 2-arm controlled clinical trial, with 3 waves of data collection. This single-blind, randomized controlled study will evaluate the efficacy of the PsyPills app in enhancing emotion regulation and reducing engagement in risky behaviors among emerging adults aged 18-29. Participants will complete demographic questions and the Suicidal Behaviors Questionnaire-Revised (SBQ-R) for safety screening. Participants will additionally complete baseline measurements for primary and secondary outcomes. Next, eligible participants will be enrolled and randomly assigned (1:1) to one of two conditions: PsyPills app (experimental group) or MoodWheel app (active control group). Among the constructs evaluated are emotion regulation difficulties; cognitive emotion regulation strategies and risky behaviors (substance use, risky sexual behavior, self-harm, aggression, disordered eating). Both intervention groups will use their assigned mobile application for a two-week period, with a minimum usage frequency of 3 sessions per week. The PsyPills app allows users to monitor and label emotions and delivers short, adaptive cognitive-behavioral interventions ("psychological pills") based on REBT principles and the JITAI framework, aiming to improve emotion regulation in real time by using rational thinking strategies to change the intensity of dysfunctional emotionality. The MoodWheel app serves as an active control, simply allowing users to monitor and label emotions without providing cognitive restructuring or feedback.

ELIGIBILITY:
Inclusion Criteria:

* High emotional regulation difficulties, but not severe (DERS total score 88-105)
* At least one risky behavior with a frequency ≥ 2 on the RBQ Frequency Scale
* Access to an Android or iOS smartphone

Exclusion Criteria:

* Diagnosed psychiatric disorders
* Suicide risk (score ≥ 7 on the Suicidal Behaviors Questionnaire-Revised, SBQ-R)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation | Baseline
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) - 36 items rated on a 5-point Likert scale (1 = almost never, 5 = almost always). Total scores range from 36 to 180, with higher scores indicating greater difficulties in emotion regulation
Change from Baseline Difficulties in Emotion Regulation at 2 weeks | Post-intervention (2 weeks)
  Change in DERS total and subscale scores, with higher decreases reflecting improved emotion regulation.
Change from Baseline Difficulties in Emotion Regulation at 1 month | Follow-up (1 month)
  Maintenance of change in DERS total and subscale scores.
Cognitive Emotion Regulation Strategies | Baseline
  Cognitive Emotion Regulation Questionnaire-romanian version (CERQ; Perte & Miclea, 2011) - 36 items across 9 subscales (e.g., reappraisal, acceptance, planning). Each subscale ranges from 4 to 20; higher scores indicate greater use of that strategy.
Change from Baseline Cognitive Emotion Regulation Strategies at 2 weeks | Post-intervention (2 weeks)
  Change in adaptive emotion regulation strategies (e.g., cognitive reappraisal, acceptance).
Change from Baseline Cognitive Emotion Regulation Strategies at 1 month | Follow-up (1 month)
  Maintenance of adaptive emotion regulation strategy use.

SECONDARY OUTCOMES:
Risky Behaviors | Baseline
  Risky Behavior Questionnaire (RBQ; Weiss et al., 2018) - self-report scale assessing the frequency and emotional context (negative and positive affect) of risky behaviors such as substance use, risky sexual behavior, self-harm, aggression, and disordered eating. Higher scores indicate higher engagement in risky behaviors.
Change from Baseline Risky Behaviors at 2 weeks | Post-intervention (2 weeks)
  Change in RBQ total and subscale scores, with reductions reflecting decreased engagement in risky behaviors.
Change from Baseline Risky Behaviors at 1 month | Follow-up (1 month)
  Maintenance of reductions in risky behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiss NH, Tull MT, Dixon-Gordon K, Gratz KL. Assessing the Negative and Positive Emotion-Dependent Nature of Risky Behaviors Among Substance Dependent Patients. Assessment. 2018 Sep;25(6):702-715. doi: 10.1177/1073191116665906. Epub 2016 Aug 30. PMID 27581175
- [Result] Perte, A. & Miclea, Mircea. (2011). The standardization of the cognitive emotion regulation questionnaire (CERQ) on Romanian population. Cognition Brain and Behavior. 15. 111-130.
- [Result] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26(1), 41-54.